CLINICAL TRIAL: NCT05591261
Title: Strong Couples Project: ePREP Nationwide Dissemination
Brief Title: Strong Couples Project: Disseminating Evidence-based Relationship Education
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21550
Record Dates: First submitted 2022-07-18; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Relationships, Marital; Relational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ePREP condition (Experimental): The ePREP program is the online version of the Prevention and Relationship Enhancement Program. It consists of 6 self-directed online sessions and accompanying homework and brief coach calls.
  Interventions: Behavioral: ePREP

INTERVENTIONS:
Behavioral: ePREP — 6-session online psychoeducational program with supporting coach calls

SUMMARY:
The current research is designed to implement and evaluate the ePREP relationship intervention with couples via the Cooperative Extension system.

DETAILED DESCRIPTION:
The objective of the research is to evaluate the effectiveness of an online intervention (ePREP) for help-seeking couples designed to promote individual and couple well-being. Newly developed online intervention programs for distressed couples have shown to be efficacious, but their overall reach to the general population remains limited. The current research is designed to implement and evaluate the ePREP relationship intervention with couples throughout the nation in a manner that allows for scalable, sustainable program delivery.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Illinois
* Married, engaged, or living with their partner for at least 6 months
* Both partners willing to participate in online relationship-focused programming

Exclusion Criteria:

* One or both partners reports sever forms of intimate partner violence occurring in the relationship

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in relationship satisfaction | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  Couple satisfaction index
Change in relationship instability | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  3 item Relationship Instability measure (from Doss et al., 2020, Journal of Consulting and Clinical Psychology
Change in partner support | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  5 item Partner Support measure (from Doss et al., 2020, Journal of Consulting and Clinical Psychology
Change in communication conflict | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  4 item communication conflict measure (from Doss et al., 2020, Journal of Consulting and Clinical Psychology
Change in relationship confidence | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  4 item relationship confidence measure (from Stanley et al., 1994)
Change in intervention-targeted behavior | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  PREP 3 keys and Couple Communal Identity (new measures created for this study)

SECONDARY OUTCOMES:
Change in partner aggression | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  7 item partner aggression (from Doss et al., 2020, Journal of Consulting and Clinical Psychology
Change in psychological distress | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  Kessler 6 item psychological distress
Change in anger | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  NIH PROMIS 5 item anger measure
Change in perceived stress | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  Cohen's 10 item perceived stress measure
Change in general health | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  Short Form-36 4 item general health perceptions
Change in insomnia | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  7 item insomnia severity index
Change in problematic alcohol use | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  Patient-Reported Outcomes Measurement Information System (PROMIS) 7 item problematic alcohol use
Change in exercise | Baseline, Within one week of program completion (~2 months post-baseline), and 6-month follow-up from baseline
  1 item exercise (Behavioral Risk Factor Surveillance System 2016 adaptation)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Extension, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No